CLINICAL TRIAL: NCT06872229
Title: How the Simultaneous or Delayed Presentation of Visual and Auditory Stimuli Affects Response Accuracy and Reaction Times in Participants With Autism Spectrum Condition (ASC) During an Association Task.
Brief Title: The Impact of Sensory Integration on Attention in Autism
Status: Recruiting | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Sponsor
Other Study IDs: CNR-IRIB-PRO-2025-002
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; autism spectrum condition; utism spectrum disorder; sensory overload; sensory processing; sensory integration
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with autism spectrum condition: Fifty ASC children with medium-high functioning, aged 4 to 12 years
  Interventions: Behavioral: Autism Spectum Conditions - intervention
- Typical development: Fifty Typical development children, aged 4 to 12 years
  Interventions: Behavioral: Typical Development - intervention

INTERVENTIONS:
Behavioral: Autism Spectum Conditions - intervention — Initially, participants will participate in a familiarization session in which they will see and hear all pairs of pictures and sounds without any associated task, thus ensuring adequate understanding of the stimuli. Next, each child will be tested for each predicted condition, receiving clear instructions on the task: they will have to indicate whether the picture and sound are related. The main task consists of presenting 40 pairs of image-sound stimuli. For each pair, participants must answer the question, "Does what you saw match what you heard?" using a keypad with a green key for "Yes" and a red key for "No." Each condition includes 10 trials, distributed randomly, with short breaks between them to keep participants focused.
  Groups: Children with autism spectrum condition
Behavioral: Typical Development - intervention — Initially, participants will participate in a familiarization session in which they will see and hear all pairs of pictures and sounds without any associated task, thus ensuring adequate understanding of the stimuli. Next, each child will be tested for each predicted condition, receiving clear instructions on the task: they will have to indicate whether the picture and sound are related. The main task consists of presenting 40 pairs of image-sound stimuli. For each pair, participants must answer the question, "Does what you saw match what you heard?" using a keypad with a green key for "Yes" and a red key for "No." Each condition includes 10 trials, distributed randomly, with short breaks between them to keep participants focused.
  Groups: Typical development

SUMMARY:
The study aims to examine how the mode of presentation of visual and auditory stimuli-separate or simultaneous-affects accuracy and reaction time in visual-auditory association in participants with Autism Spectrum Condition (ASC) compared to neurotypical individuals. The study aims to evaluate whether sensory overlap (simultaneous stimuli) increases cognitive load and decreases performance, while stimulus separation (separate presentation of visual and auditory stimuli) may facilitate processing and improve performance, especially in participants with ASC. Participants will be divided into two main groups: the first consisting of individuals with ASD and the second of neurotypical individuals. Each group will be exposed to two modes of stimulus presentation: simultaneous mode, in which visual and auditory stimuli are presented at the same time, and separate mode, in which visual and auditory stimuli are presented separately with a time interval between each. Participants will be required to complete visual-auditory association tasks. In addition to assessment of reaction time and accuracy, psychophysiological parameters will be recorded to measure cognitive load and physiological reaction to stimuli. The main hypotheses are that the simultaneous presentation of visual and auditory stimuli will increase cognitive load and reduce accuracy and reaction time in individuals with ASC, while the separate mode will improve performance, especially in the group with ASC. This study could provide important insights into how stimulus presentation mode affects learning and performance in participants with ASC, suggesting that stimulus separation could be a useful strategy for optimizing sensory processing and improving learning in educational and therapeutic settings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism
* QI ≥ 80

Exclusion Criteria:

* significant hearing or visual impairments
* presence of other medical disorders
* history of psychiatric diagnosis

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifty children with Autism Spectrum Condition (ASC) and fifty typically developing (TD) children will participate in the study. The children with ASC will be recruited and tested at the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina. To be included in the study the child needs to have an ASD diagnosis based on the DSM-5 criteria from a licensed clinical child neuropsychiatrist but no established intellectual disability (ID) diagnosis. The TD children will recruit through advertisements in schools located close to the Institute. Informed consent will be obtained from all subjects involved in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | The session needs approximately 50 minutes to complete
  Accuracy will be calculated for each answer. The percentage of correct answers for the 50 tests provided will be calculated
Reaction time | The session needs approximately 50 minutes to complete
  The time between delivery and the response given by the child for each task will be calculated in seconds (s)
Heart rate variability | The heart rate variability will be measured throughout the session (approximately 50 minutes)
  The electrical activity of the heart will be measured with a heart rate sensor with a chest strap

SECONDARY OUTCOMES:
Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) | The evaluation session will be scheduled pre-intervention. The test needs approximately 65-80 minutes
  Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) is a clinical tool for assessing the cognitive abilities of children and young people between the ages of 6 years and 16 years and 11 months.
The Sensory Profile 2 | The evaluation session will be scheduled pre-intervention. The test needs approximately 5-15 minutes
  The Sensory Profile 2 is a standardized battery of self-administered caregiver questionnaires documenting the sensory processing patterns of children from birth to 14.11 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, ME, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevenson RA, Siemann JK, Woynaroski TG, Schneider BC, Eberly HE, Camarata SM, Wallace MT. Evidence for diminished multisensory integration in autism spectrum disorders. J Autism Dev Disord. 2014 Dec;44(12):3161-7. doi: 10.1007/s10803-014-2179-6. PMID 25022248
- [Background] Noel JP, De Niear MA, Stevenson R, Alais D, Wallace MT. Atypical rapid audio-visual temporal recalibration in autism spectrum disorders. Autism Res. 2017 Jan;10(1):121-129. doi: 10.1002/aur.1633. Epub 2016 May 9. PMID 27156926
- [Background] Font-Alaminos M, Cornella M, Costa-Faidella J, Hervas A, Leung S, Rueda I, Escera C. Increased subcortical neural responses to repeating auditory stimulation in children with autism spectrum disorder. Biol Psychol. 2020 Jan;149:107807. doi: 10.1016/j.biopsycho.2019.107807. Epub 2019 Nov 3. PMID 31693923
- [Background] Zhou HY, Yang HX, Shi LJ, Lui SSY, Cheung EFC, Chan RCK. Correlations Between Audiovisual Temporal Processing and Sensory Responsiveness in Adolescents with Autistic Traits. J Autism Dev Disord. 2021 Jul;51(7):2450-2460. doi: 10.1007/s10803-020-04724-9. PMID 32978707